CLINICAL TRIAL: NCT05031156
Title: Effect of Mandibular Immediately Loaded, Screw-retained Splinted and Non-splinted OT Bridge Implant Restoration on Bone Height Changes of Completely Edentulous Patients (A Randomized Clinical Trial)
Brief Title: Splinted and Unsplinted OT Bridge Systems in Screw Retained Implant Restoration
Acronym: OTBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, tasneem gamal youssef el mashad, Assistant lecturer of Prosthodontics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OTBridge
Record Dates: First submitted 2021-08-29; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Evaluate the Immediate Loading Implants in All on 4 Cases Using Conversion Denture and OT Bridge System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-splinting of OT Bridge system (Active Comparator): Leaving the dental implants abutments solitary followed by denture pick up
  Interventions: Procedure: Splinting of OT Bridge system
- splinting of OT Bridge (Experimental): Splinting of implants abutments using titanium wire then followed by denture pick up
  Interventions: Procedure: Splinting of OT Bridge system

INTERVENTIONS:
Procedure: Splinting of OT Bridge system — splinting of implant abutment using titanium wire followed by pick up using the patient's denture

SUMMARY:
Evaluation of Bone level changes around dental implants in All on 4 cases with immediate loading using conversion denture and OT Bridge system either splinted or not

ELIGIBILITY:
Inclusion Criteria:

* Any completely edentulous patient (mandible) with an old satisfactory denture requiring an implant-supported restoration.
* Patients aged from 40 to 70, able to sign an informed consent will be considered eligible for this trial.
* Implant sites must allow the placement of four implants.
* Non- heavy Smokers will be included (smoking up to 10 cigarettes/day)
* In case of post-extractive sites, they must have been healed for at least 3-month before being treated in the study.
* Patients with no systemic condition that may interfere with implant placement (e.g., Immunosuppressed or immunocompromised patients, patients under treatment of intravenous amino-bisphosphonates)

Exclusion Criteria:

* - Patients with poor oral hygiene and motivation.
* Pregnancy or nursing.
* Drug abusers.
* Psychiatric problems or unrealistic expectations.
* Patients with infection and or inflammation in the area intended for implant placement.
* Patients participating in other studies, if the present protocol cannot be properly adhered to.
* Patients with signs of hyperactive muscles.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-07 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone loss | 3 monts
  Measures the changes around the dental implants along the healing period using paralleling technique radiograph and DIGORA system

SECONDARY OUTCOMES:
Early implant failure | 3 months
  not fulfilling one of Alberksston implant success criteria

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem El Mashad, Principal Investigator — Cairo University